CLINICAL TRIAL: NCT05576675
Title: Patient-controlled Intravenous Analgesia Combined With Different Opioid Receptors for Gastrointestinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xijingHospital
Record Dates: First submitted 2022-09-01; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-08

CONDITIONS: Gastrointestinal Surgery
Keywords: patient-controlled intravenous analgesia; gastrointestinal surgery
MeSH Terms: interventions — Sufentanil; Nalbuphine; Hydromorphone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SN group (Experimental): sufentanil 100 μ g + nalbuphine 40 mg
  Interventions: Drug: sufentanil + nalbuphine
- HN group (Experimental): hydromorphone 10 mg+ nalbuphine 40 mg
  Interventions: Drug: hydromorphone + nalbuphine
- S group (Experimental): sufentanil 200 μ g,
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: sufentanil + nalbuphine — sufentanil 100 μ g + nalbuphine 40 mg
  Arms: SN group
Drug: Sufentanil — sufentanil 200 μ g
  Arms: S group
Drug: hydromorphone + nalbuphine — hydromorphone 10 mg+ nalbuphine 40 mg
  Arms: HN group

SUMMARY:
Objective To evaluate the effect of patient-controlled intravenous analgesia combined with different opioid receptors for gastrointestinal surgery. Methods A total of 4342 patients who underwent gastrointestinal postoperative analgesia in the first affiliated Hospital of Air Force military Medical University from May 2018 to March 2022 were collected retrospectively. The patient-controlled intravenous analgesia regimen in this study was composed of different opioid receptor drugs：sufentanil combined with nalbuphine group (SN group) and Hydromorphone combined with nalbuphine group (HN group) and single opioid receptor group: sufentanil group (S group). SN group ,HN group and S group were treated with sufentanil 100 μ g + nalbuphine 40 mg, hydromorphone 10 mg+ nalbuphine 40 mg, sufentanil 200 μ g, diluted to 100 ml, background dose 1 ml/h, PCA dose 0.5 ml, locking time 10 min. The demographic data of the three groups were collected, the number of patients with insufficient static and dynamic analgesia (VAS ≥ 4) at 24 and 48 hours after operation, the adverse reactions at 24 and 48 hours after operation, the first exhaust time and the first ambulation time were collected, evaluate the analgesic effect of combination of different opioid receptor drugs and single opioid receptor drugs in PCIA after gastrointestinal surgery.

DETAILED DESCRIPTION:
Control group：S group Test group：SN group and HN group Observation index：the number of patients with insufficient static and dynamic analgesia (VAS ≥ 4) at 24 and 48 hours after operation, the adverse reactions（drowsiness, nausea and vomiting, respiratory depression, dizziness） at 24 and 48 hours after operation, the first exhaust time and the first ambulation time were collected

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years ,there is no gender limit，ASA grade Ⅰ-Ⅱ

Exclusion Criteria:

* BMI > 35 kg/m2, history of upper abdominal surgery, history of analgesic or hormone use before operation, history of depression or chronic pain before operation, infection before operation and ICU after operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4342 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
the incidence of insufficient static and dynamic analgesia dynamic analgesia | 24 hours after operation
  VAS ≥ 4
the incidence of insufficient static and dynamic analgesia dynamic analgesia | 48 hours after operation
  VAS ≥ 4

SECONDARY OUTCOMES:
the incidence of adverse reactions | 24 hours after operation
  dizziness, nausea and vomiting
the incidence of adverse reactions | 48 hours after operation
  dizziness, nausea and vomiting

OTHER OUTCOMES:
first exhaust time | immediately after operation
  first exhaust time
first ambulation time | immediately after operation
  first ambulation time

CONTACTS AND LOCATIONS:
Overall Officials: Yan LI, Study Chair — The First Affiliated Hospital of the Air Force Medical Universtiy; jing LIN, Study Chair — The First Affiliated Hospital of the Air Force Medical Universtiy
Locations (1):
- YANLI, XIan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No